CLINICAL TRIAL: NCT00610324
Title: Effect of Oral Decontamination Using Chlorhexidine or Potassium Permanganate in ICU Patients: an Open-Labelled Randomized Controlled Trial
Brief Title: Effect of Oral Decontamination Using Chlorhexidine or Potassium Permanganate in ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Memorial Hospital (Other)
Responsible Party: Dr Dilip Karnad, Professor of Medicine, K E M Hospital, Mumbai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DRK-CHEX
Record Dates: First submitted 2008-01-16; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Nosocomial Pneumonia; Healthcare-Associated Pneumonia; Aspiration Pneumonia; Ventilator-Associated Pneumonia
Keywords: oropharyngeal cleansing; oral decontamination; oropharyngeal bacterial flora; oropharyngeal colonization; critical illness; mechanical ventilation; tracheal intubation; prophylaxis
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Aspiration; Pneumonia, Ventilator-Associated; Critical Illness | interventions — chlorhexidine gluconate; Potassium Permanganate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Twice-daily oropharyngeal cleansing with 0.2% Chlorhexidine gluconate
  Interventions: Drug: Chlorhexidine gluconate
- 2 (Active Comparator): Twice-daily oropharyngeal cleansing with 0.01% Potassium permanganate
  Interventions: Drug: Potassium permanganate

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Twice-daily oropharyngeal cleansing with 0.2% Chlorhexidine gluconate
  Arms: 1
Drug: Potassium permanganate — Twice-daily oropharyngeal cleansing with 0.01% Potassium permanganate
  Arms: 2

SUMMARY:
Oropharyngeal bacteria play an important role in the pathogenesis of nosocomial pneumonia in critically ill patients. Oral cleansing with chlorhexidine has been shown to decrease incidence of pneumonia in patients undergoing open heart surgery. Its role in critically ill general ICU patients is not yet proven. The present study proposes to study the effectiveness of twice-daily oral cleansing with 0.2% chlorhexidine solution on the incidence of nosocomial pneumonia in ICU patients admitted to a single intensive care unit of an Indian public hospital

DETAILED DESCRIPTION:
Nosocomial pneumonia is common in intensive care units (ICU) patients and is associated with increase in mortality rates by 24% to 76% in various studies. Interventions that effectively prevent nosocomial pneumonia are strategically important in order to reduce morbidity, mortality and healthcare costs. Colonization of the pharynx has been implicated as the reservoirs for pathogens causing nosocomial pneumonia and interventions like selective digestive decontamination have been tried to control this source of infection. Recently, colonization of the dental plaque by aerobic organisms with subsequent aspiration into the lower respiratory tract has received attention. Previous smaller studies using antiseptic agents to sterilize dental plaques in patients at risk of pneumonia have shown conflicting results. The present study aims to determine whether twice daily oral cleansing with 0.2% chlorhexidine reduces the incidence of nosocomial pneumonia in patients staying in the ICU for >48 hours.

After obtaining informed consent, subjects would be randomized to treatment with either 0.2% chlorhexidine gluconate (CHG) solution or 0.01% potassium permanganate solution (PP) (Control Group), as per the protocol approved by the Institutional Ethics Committee. At baseline, the parameters which would be noted are: age, sex, surgical or non-surgical status, immunosuppression, chronic ailments, smoking and alcohol consumption, Glasgow coma scale score (GCS), laboratory parameters and blood gas analysis. All subjects would be followed up daily and the GCS, presence of nasogastric tube (feeds), endotracheal tube, tracheostomy, ventilator, central venous and urinary catheterization, anti-stress ulcer prophylaxis and prior antibiotic use will be noted. Presence or absence of nosocomial pneumonia would also be noted daily. Lower respiratory secretions would be obtained by the protected non-bronchoscopic mini-BAL technique in order to identify the causative organisms. All the subjects will be followed up daily until discharge from the ICU or death.

Primary outcome variable was the development of nosocomial pneumonia during the ICU stay. Secondary outcome variables were hospital mortality, length of ICU stay.

A total of 506 patients will have to be studied (approximately 253 patients in each treatment group). This study will have a statistical power of 75% to detect a 50% reduction in the incidence of nosocomial pneumonia in the intervention group with a 95% level of confidence assuming that incidence of pneumonia in the control group is 16%.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the medical intensive care unit and are expected to stay in ICU for > 48 hours

Exclusion Criteria:

* Pregnant women
* Patients with nosocomial pneumonia at time of ICU admission
* Patients with community-acquired pneumonia at time of ICU admission
* Patients in whom oropharyngeal cleansing is contra-indicated

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2004-05; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Development of nosocomial pneumonia | During hospital stay

SECONDARY OUTCOMES:
In-hospital mortality | During hospital stay
Length of ICU stay (days) | Till discharge from ICU or death

CONTACTS AND LOCATIONS:
Overall Officials: Dilip R Karnad, MD,FACP,FRCP, Principal Investigator — Professor of Medicine, K E M Hospital, Parel, Mumbai 400012, India
Locations (1):
- Medical-Neuro Intensive Care Unit, K E M Hospital, Parel, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Abele-Horn M, Dauber A, Bauernfeind A, Russwurm W, Seyfarth-Metzger I, Gleich P, Ruckdeschel G. Decrease in nosocomial pneumonia in ventilated patients by selective oropharyngeal decontamination (SOD). Intensive Care Med. 1997 Feb;23(2):187-95. doi: 10.1007/s001340050314. PMID 9069004
- [Background] DeRiso AJ 2nd, Ladowski JS, Dillon TA, Justice JW, Peterson AC. Chlorhexidine gluconate 0.12% oral rinse reduces the incidence of total nosocomial respiratory infection and nonprophylactic systemic antibiotic use in patients undergoing heart surgery. Chest. 1996 Jun;109(6):1556-61. doi: 10.1378/chest.109.6.1556. PMID 8769511
- [Background] Fourrier F, Cau-Pottier E, Boutigny H, Roussel-Delvallez M, Jourdain M, Chopin C. Effects of dental plaque antiseptic decontamination on bacterial colonization and nosocomial infections in critically ill patients. Intensive Care Med. 2000 Sep;26(9):1239-47. doi: 10.1007/s001340000585. PMID 11089748
- [Background] Francis JR, Hunter B, Addy M. A comparison of three delivery methods of chlorhexidine in handicapped children. I. Effects on plaque, gingivitis, and toothstaining. J Periodontol. 1987 Jul;58(7):451-5. doi: 10.1902/jop.1987.58.7.451. PMID 2957488